CLINICAL TRIAL: NCT06345170
Title: Investigation the Effect of the Social-Communication Area Developmental Screening Test for Infants and Young Children Training Program Applied in Addition to the DIR/Floortime™ Therapy Program in Children with Developmental Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Hikmet Ucgun, Assistant Professor, Biruni University
Allocation: Not Applicable | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: buhucgun05
Record Dates: First submitted 2024-03-28; First posted 2024-04-03 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2024-05

CONDITIONS: Children with Developmental Risk
Keywords: Children; Developmental Risk; DIR/Floortime; Social-Communication Area Developmental Screening Test for Infants and Young Children (SCASI); Social Communication
MeSH Terms: conditions — Communication

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): The group in which the Social-Communication Area Developmental Screening Test for Infants and Young Children (SCASI) training program will be applied in addition to the DIR/Floortime™ therapy program
  Interventions: Other: The DIR/Floortime™ Therapy Program; Other: The Social-Communication Area Developmental Screening Test for Infants and Young Children (SCASI) Training Program
- Control Group (Active Comparator): The group in which the DIR/Floortime™ therapy program will be applied
  Interventions: Other: The DIR/Floortime™ Therapy Program

INTERVENTIONS:
Other: The DIR/Floortime™ Therapy Program — The DIR/Floortime™ therapy program will be applied by the therapist in the clinic for 50 minutes, 2 days a week for 12 weeks
Other: The Social-Communication Area Developmental Screening Test for Infants and Young Children (SCASI) Training Program — The Social-Communication Area Developmental Screening Test for Infants and Young Children (SCASI) Training Program will be applied by the parents at home, 2 days a week, for an average of 30 minutes a day, for 12 weeks
  Arms: Intervention Group

SUMMARY:
The term "developmental risk" is used as a general term for developmental delays observed in infancy and early childhood. Developmental delay refers to the delay in children reaching developmental milestones compared to their peers. The DIR/Floortime™ therapy program is an approach that uses play as a therapeutic tool, emphasising the importance of interaction involving affect and excitement in a child's development. DIR/Floortime™ therapy program aims to support the child's development with a family-centred perspective by evaluating the child and the family together. DIR/Floortime™ therapy program is known to contribute to the functional and emotional development of children and the development of parenting skills of caregivers. The Social-Communication Area Developmental Screening Test for Infants and Young Children (SCASI) is a parent-reported developmental screening test that aims to identify 'delays' in the social communication area skills of infants and children. The SCASI training program is a training program for children and parents developed on the basis of this screening test, which includes targeted activities to support the development process according to the child's developmental level. To the best of our knowledge, there is no study investigating the effect of the SCASI training program applied in addition to the DIR/Floortime™ therapy program in children with risky development. The aim of the study is to examine the effect of the SCASI training program applied in addition to the DIR/Floortime™ therapy program in children with risky development. A total of 34 children with developmental risk between the ages of 1 and 3 will included in the study. Participants will randomly divided into two groups: control group (n=17) in which the DIR/Floortime™ therapy program will be applied and intervention group (n=17) in which the SCASI training program will be applied in addition to the DIR/Floortime™ therapy program. The DIR/Floortime™ therapy program will be applied by the therapist in the clinic for 50 minutes, 2 days a week for 12 weeks, and the SCASI training program will be applied by the parents at home, 2 days a week, for an average of 30 minutes a day, for 12 weeks. Demographic and clinic informations, SCASI test, Age and Stages Questionnarie (ASQ), Age and Stages Questionnaires: Social-Emotional (ASQ-SE) and Brief Infant and Toddler Social Emotional Assessment (BITSEA) will be used as outcome measures in the study.

ELIGIBILITY:
Inclusion Criteria:

* The child is between 1-3 years old
* The language of the parents and the child is Turkish
* Assessment of SİATT pre-test result as "developmental risk"
* Parents' willingness to participate in the study

Exclusion Criteria:

* Any cognitive impairment in the parents that may interfere with communication
* Illiteracy of parents
* The child has orthopedic, neurological disability(s) other than developmental risk

Ages: 1 Year to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2022-10-30 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
The Social-Communication Area Developmental Screening Test for Infants and Young Children (SCASI) | 12 weeks
Age and Stages Questionnarie (ASQ) | 12 weeks
Age and Stages Questionnaires: Social-Emotional (ASQ-SE) | 12 weeks
Brief Infant and Toddler Social Emotional Assessment (BITSEA) | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Biruni University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No